CLINICAL TRIAL: NCT00637767
Title: A Randomised Phase II Clinical Trial Using Targeted Radiotherapy Delivered by an Yttrium-90 Radio-Labelled Anti-CD66 Monoclonal Antibody With High Dose Melphalan Compared to Melphalan Alone, Prior to Autologous Stem Cell Transplantation for Multiple Myeloma
Brief Title: High-Dose Melphalan With or Without Radiolabeled Monoclonal Antibody in Treating Patients With Multiple Myeloma Undergoing an Autologous Stem Cell Transplant
Acronym: AntiCD-66
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: University of Southampton (Other)
Collaborators: NIHR Clinical Research Facility, University Hospital Southampton NHS Foundation Trust (Unknown); European Federation of Pharmaceutical Industries and Associations (Unknown); Bill and Melinda Gates Foundation (Other); The Periscope Consortium (Unknown); Q-Biologicals NV (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000588063; 2006-003424-12 (EudraCT Number); EU-20820 (Other: EU)
Record Dates: First submitted 2008-03-14; First posted 2008-03-18 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Melphalan; BW 250 183

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radio-labelled anti-CD66 monoclonal antibody (Experimental): Up to 4mg radio-labelled anti-CD66 monoclonal antibody. Plus standard treatment
  Interventions: Drug: melphalan; Procedure: autologous hematopoietic stem cell transplantation; Radiation: yttrium Y 90 anti-CD66 monoclonal antibody BW 250/183
- No IMP - standard treatment (Active Comparator): No IMP - standard treatment
  Interventions: Drug: melphalan; Procedure: autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: melphalan
Procedure: autologous hematopoietic stem cell transplantation
Radiation: yttrium Y 90 anti-CD66 monoclonal antibody BW 250/183
  Arms: radio-labelled anti-CD66 monoclonal antibody

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiolabeled monoclonal antibodies can find cancer cells and carry cancer-killing substances to them without harming normal cells. A stem cell transplant using stem cells from the patient may be able to replace blood-forming cells that were destroyed by the chemotherapy and radiolabeled monoclonal antibody.

PURPOSE: This randomized phase II trial is studying how well high-dose melphalan works when given with or without radiolabeled monoclonal antibody in treating patients with multiple myeloma undergoing an autologous stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of high-dose melphalan (200mg/m²) in combination with targeted radiotherapy delivered by yttrium Y 90 anti-CD66 monoclonal antibody BW250/183, in terms of disease response (complete remission rate and change in serum free light chain level before and after treatment with yttrium Y 90 anti-CD66 monoclonal antibody BW250/183), in patients undergoing autologous hematopoietic stem cell transplantation for multiple myeloma.

Secondary

* To determine the toxicity profile of yttrium Y 90 anti-CD66 monoclonal antibody BW250/183 in the context of autologous hematopoietic stem cell transplantation.
* To determine the effect of targeted radiotherapy on other parameters of disease response, in terms of proportion of patients with partial remission, stable disease, and progressive disease, remission duration (time to disease progression), and overall survival.
* To determine the effect of targeted radiotherapy on engraftment when used in combination with high-dose melphalan in patients undergoing autologous hematopoietic stem cell transplantation for multiple myeloma.
* To investigate the pharmacokinetic behavior of indium In 111 anti-CD66 monoclonal antibody BW250/183 (used for dosimetry).
* To continue to develop a dosimetry model based on single-photon emission computed tomography (SPECT) and whole body gamma camera imaging following administration of the radiolabeled anti-CD66 monoclonal antibody (in a subset of patients at the Southampton site only).
* To assess the proportion of patients who form human anti-murine antibodies (HAMA) after treatment with targeted radiotherapy in the context of an autologous hematopoietic stem cell transplantation.

OUTLINE: This is a multicenter study. Patients are stratified according to disease risk group (low risk [beta-2 microglobulin and C-reactive protein < 6 or either beta-2 microglobulin or C-reactive protein ≥ 6] vs high risk [both beta-2 microglobulin and C-reactive protein ≥ 6]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive a dosimetry dose of indium In 111 anti-CD66 monoclonal antibody BW250/183 IV on day 1 and undergo gamma camera imaging and serial blood samples on days 1-5. Patients then receive a therapeutic dose of yttrium Y 90 anti-CD66 monoclonal antibody BW250/183 IV once between days 9 and 16 and high-dose melphalan IV on day 28. Patients then undergo autologous hematopoietic stem cell transplantation (HSCT) on day 30.
* Arm II: Patients receive high-dose melphalan IV on day 1. Patients then undergo autologous HSCT on day 3.

Patients in arm I undergo blood sample collection periodically for pharmacokinetic and pharmacodynamic studies and analysis of human anti-murine antibody (HAMA) status.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven multiple myeloma (MM)
* Scheduled to undergo autologous hematopoietic stem cell transplantation (HSCT) as consolidation treatment for MM

  * Must have sufficient CD34-positive stem cells (≥ 4 x 10^6 cells per kg body weight) in cryo-storage for two autologous HSCTs
* In partial remission (PR) after prior chemotherapy but before priming therapy for stem cell mobilization

  * Patients in complete remission (CR) after prior chemotherapy are not eligible
* Bone marrow cellularity ≥ 20%

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy ≥ 24 weeks
* Hemoglobin ≥ 9.0 g/dL
* Neutrophils ≥ 1,500/mm³
* Platelets ≥ 50,000/mm³
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and/or AST ≤ 2.5 times ULN
* Creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use effective contraception for 4 weeks prior to, during, and for 6 months after completion of study treatment
* Fertile male patients must use effective contraception during and for 6 months after completion of study treatment
* Able to cooperate with study treatment and follow up
* Human anti-mouse antibody (HAMA) negative
* No active uncontrolled infection
* No high-risk non-malignant systemic disease
* No other condition, that in the investigator's opinion, would make the patient an unsuitable candidate for the study
* No known HIV or hepatitis B or C seropositivity
* No history of allergy, including an allergy to rodents or rodent proteins
* No history of eczema or asthma
* No history of New York Heart Association (NYHA) class III or IV cardiac disease
* No congestive heart failure

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy

  * Alopecia or certain grade 1 toxicities allowed
* More than 4 weeks since prior radiotherapy (except for localized pain control), endocrine therapy, or immunotherapy
* More than 4 weeks since prior and no other concurrent chemotherapy for the underlying hematological condition, except for the following:

  * Cyclophosphamide as priming for stem cell harvest
  * Thalidomide
* More than 3 weeks since prior major thoracic and/or abdominal surgery and recovered
* No prior high-dose therapy and autologous HSCT
* Concurrent radiotherapy allowed for the control of bone pain

  * The irradiated lesions are not used for response evaluation
* No other concurrent anti-cancer therapy or investigational drugs during transplantation conditioning

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2013-10-31 (Actual); Study Completion 2013-10-31 (Actual)

PRIMARY OUTCOMES:
Remission status pre- and post-transplantation, specifically the number of patients who achieve complete remission, as measured by the European Blood and Marrow Transplantation Organization Response Criteria | end of study

SECONDARY OUTCOMES:
Disease response, as measured by changes in serum free light chains (in those patients with serum free light chains that are informative) | end of study
Disease response, including the proportion of patients with partial remission, stable disease, and progressive disease and remission duration (time to disease progression) | end of study
Engraftment quality, as measured by time to recovery of peripheral blood neutrophils to > 500/mm³ and platelets > 50, 000/mm³ and duration of recovery for > 180 days post-transplantation | end of study
Treatment-related mortality | end of study
Overall survival | end of study
Toxicity profile of yttrium Y 90 anti-CD66 monoclonal antibody BW250/183 in the context of autologous stem cell transplantation | end of study
Pharmacokinetics of indium In 111 anti-CD66 monoclonal antibody BW250/183 as measured by serial blood samples and serial planar and single-photon emission computed tomography (SPECT) gamma camera imaging of selected organs | end of study
Development of a dosimetry model based on SPECT and whole body gamma camera imaging | end of study
Proportion of patients who form human anti-murine antibodies (HAMA) after treatment with targeted radiotherapy in the context of an autologous hematopoietic stem cell transplantation | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Kim Orchard, MD, Study Chair — University Hospital Southampton NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Saint Bartholomew's Hospital, London, England
  - Southampton General Hospital, Southampton, England